CLINICAL TRIAL: NCT04064294
Title: Preventing Levodopa Induced Dyskinesia in Parkinson's Disease With Statins
Brief Title: Preventing Levodopa Induced Dyskinesia in Parkinson's Disease With HMG-CoA Reductase Inhibitors
Acronym: STAT-PD
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: NURE-004-18S; 17302 (Other Grant/Funding Number: Oregon Health and Science University); 3869 (Other: VA Portland Health Care System); 5273 (Other: Oregon Clinical & Translational Research Institute); 1635227 (Other: VA Portland Health Care System (IRBNet))
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Dyskinesia, Drug-Induced
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced | interventions — Infusions, Intravenous; Levodopa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Statin Before Levodopa: Historical use of a statin BEFORE beginning levodopa
  Interventions: Drug: Intravenous Infusion
- Statin After Levodopa: Historical use of a statin AFTER beginning levodopa
  Interventions: Drug: Intravenous Infusion
- No Statin: No historical use of a statin
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion — Intravenous levodopa given 1.0 to 1.5 mg/kg/hr from 0930 - 1130 on a single visit day.
  Other Names: levodopa

SUMMARY:
In this study, the investigators will examine the association of statin use and dyskinesia in a convenience sample Parkinson's disease patients in the Veterans Administration Health Care System.

DETAILED DESCRIPTION:
Long term treatment with levodopa, the gold standard treatment of Parkinson's disease (PD), can lead to the development of abnormal involuntary movements called levodopa induced dyskinesia (LID). The severity of LID can range from mild to severely debilitating. A majority of PD patients will develop LID in their treatment life-time. In a recent study of the MPTP monkey model of PD, statin use was found to reduce LID (45%) without a worsening of Parkinsonism symptoms1. Another study showed rats treated with lovastatin prior to and with initiation of levodopa after substantia nigra lesioning showed dramatically less LID evolution compared to animals without lovastatin exposure2. In this study, the investigators will examine the association of statin use and dyskinesia in a convenience sample Parkinson's disease patients in the Veterans Administration Health Care System. This study is a retrospective three cohort design and will compare statin exposure BEFORE beginning LD, versus statin exposure AFTER LD is begun, versus NO statin exposure in PD subjects controlling for disease characteristics (severity), gender, and total LD exposure The primary endpoint is the severity of LID between the groups after years of opportunity to develop LID. Levodopa-Induced dyskinesia is a major cause of reduced quality of life for Veterans with PD and, in some cases, leads to costly surgical interventions. This project examines the impact of statin use on the presence of LID, and could lead to a future intervention trial. The reduction, delayed onset, or elimination of LID could improve the quality of life of many Veterans nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease
* Age diagnosed with Parkinson's Disease greater than or equal to 50 years
* Treatment with levodopa greater than or equal to 5 years

Exclusion Criteria:

* Deep Brain stimulation
* Unable to stand for 1 minute intervals, or sensory deficits in the feet
* Significant cognitive impairment as measured by the Montreal Cognitive Assessment score of < 18
* Subjects with unstable medical or psychiatric conditions (including hallucinations).
* History of unstable medical conditions (i.e. active cardiac disease, recent unwellness, surgery etc.)
* Current use of drugs that may affect parkinsonism or dyskinesia:

  * dopamine receptor blocking medications
  * depakote
  * lithium
  * amiodarone
  * tetrabenazine
  * metoclopramide
  * dronabinol
  * and illicit drugs such as marijuana (THC)
  * cocaine
  * methamphetamine
  * Statins other than simvastatin or lovastatin, atorvastatin ie. fluvastatin (rationale is that while all other statins are thought to not cross the blood brain barrier well, the central nervous system penetrating nature of others is not perfectly clear and could confound results)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Anne Chung, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (3):
- United States (3):
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data be available (including data dictionaries). Individual participant data that underlie the results reported the resultant article, after deidentification (text, tables, figures, and appendices). In addition to data, the study protocol and the informed consent form (ICF) will be provided. Data will be available beginning 6 months and ending 2 years following article publication. Data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Data will be released to achieve aims in the approved proposal or for individual participant data meta-analysis. Proposals may be submitted up to 24 months following article publication. After 24 months the data will be available in the investigators' VA'S data repository but without investigator support other than deposited metadata.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 5 months and ending 2 years following article publication.
Access Criteria: Data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
URL: http://www.parkinsons.va.gov/northwest/

REFERENCES:
- [Background] Obeso JA, Rodriguez-Oroz MC, Rodriguez M, DeLong MR, Olanow CW. Pathophysiology of levodopa-induced dyskinesias in Parkinson's disease: problems with the current model. Ann Neurol. 2000 Apr;47(4 Suppl 1):S22-32; discussion S32-4. PMID 10762129
- [Background] Tison F, Negre-Pages L, Meissner WG, Dupouy S, Li Q, Thiolat ML, Thiollier T, Galitzky M, Ory-Magne F, Milhet A, Marquine L, Spampinato U, Rascol O, Bezard E. Simvastatin decreases levodopa-induced dyskinesia in monkeys, but not in a randomized, placebo-controlled, multiple cross-over ("n-of-1") exploratory trial of simvastatin against levodopa-induced dyskinesia in Parkinson's disease patients. Parkinsonism Relat Disord. 2013 Apr;19(4):416-21. doi: 10.1016/j.parkreldis.2012.12.003. Epub 2012 Dec 31. PMID 23283428
- [Background] Pavon N, Martin AB, Mendialdua A, Moratalla R. ERK phosphorylation and FosB expression are associated with L-DOPA-induced dyskinesia in hemiparkinsonian mice. Biol Psychiatry. 2006 Jan 1;59(1):64-74. doi: 10.1016/j.biopsych.2005.05.044. Epub 2005 Sep 1. PMID 16139809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 2 academic medical centers and 1 Veterans administration hospital between July 2019 and March 2024. The first participant was enrolled on August 2019 and the last participant was enrolled in February 2024.
Pre-assignment Details: Of the 93 consented participants, 5 did not meet inclusion criteria. Of the 88 enrolled participants, 8 did not complete the intravenous levodopa day visit - 1 was cancelled and did not want to reschedule due to COVID-19 restrictions, 2 past away in the time between the screen and the day visit, 1 no-showed for the day visit, 2 were lost to follow-up, and 2 indicated that they were too busy to attend a full day visit. 80 participants attended the day visit.
Period: Overall Study
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
Started | 29 | 16 | 35
Completed | 28 | 16 | 35
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant experienced nausea/vomiting, the infusion was discontinued and all study related data gathering was discontinued. Dropped from the analysis due to not enough information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin | Total
Number analyzed (Participants) | 28 | 16 | 35 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (4.3) | 72.0 (7.0) | 70.6 (6.4) | 72.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9 | 18
  Male | 21 | 14 | 26 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 16 | 34 | 77
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 28 | 16 | 34 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Pacific Northwest - United States
  Participants
    United States | 28 | 16 | 35 | 79
Education [Mean (Standard Deviation); unit: years] | 16.6 (2.6) | 16.9 (3.0) | 16.4 (3.0) | 16.5 (2.8)
Age at Parkinson's Diagnosis [Mean (Standard Deviation); unit: years] — Date of Parkinson's Diagnosis - Date of Birth in years.
  years | 66.2 (5.7) | 59.4 (7.2) | 60.7 (6.4) | 62.3 (6.9)
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: years] — Date of Screening Visit - Date of Parkinson's Diagnosis in years.
  years | 8.9 (3.0) | 12.7 (5.0) | 9.9 (3.7) | 10.1 (4.0)
Hoehn & Yahr Rating [Mean (Standard Deviation); unit: units on a scale] — This is an objective staging scale for rating the clinical functioning of Parkinson's disease patients, combining functional deficits (disability) and objective signs (impairment). This staging scale is commonly used in both research settings and clinical practice. The Hoehn & Yahr is an ordinal scale ranging from 0 (no signs of disease) to 5 (wheelchair bound/bedridden). The modified version of the scale includes increments of 0.5.
  units on a scale | 2.8 (0.8) | 2.6 (0.7) | 2.5 (0.7) | 2.6 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Peak Unified Dyskinesia Rating Score (UDysRS)
Description: The Unified Dyskinesia Rating Scale (UDysRS) combines patient, caregiver, and treating physician perspectives on both historical (Parts 1 & 2) and objective (Part 3 & 4) assessments of dyskinesia and dystonia. The historical portion and the objective ratings are added together to form total score ranging from 0 to 104 with higher scores indicating more severe dyskinesia.
Time Frame: 11:00 am
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
Number analyzed (Participants) | 28 | 16 | 35
score on a scale | 10.9 (10.5) | 10.8 (11.1) | 13.2 (10.9)
Statistical Analysis 1: Comparison: No Statin; Test type: Superiority; p = 0.63, ANOVA — the threshold for statistical significance was p = 0.05; degrees of freedom = 78

2. Secondary Outcome: Peak Unified Dyskinesia Rating Scale - Objective Measures
Description: The Unified Dyskinesia Rating Scale (UDysRS) objective (Part 3 & 4) assessments of dyskinesia and dystonia. The objective ratings are added together to form total score ranging from 0 to 44 with higher scores indicating more severe dyskinesia.
Time Frame: 11:00 am
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
Number analyzed (Participants) | 28 | 16 | 35
score on a scale | 5.5 (5.1) | 3.8 (4.2) | 6.8 (4.3)
Statistical Analysis 1: Comparison: No Statin; Test type: Superiority; p = 0.09, ANOVA — the threshold for statistical significance was p = 0.05; degrees of freedom = 78

3. Secondary Outcome: Presence/Absence of Levodopa-induced Dyskinesia (LID).
Description: Any score greater than or equal to 1 on the Clinical Dyskinesia Rating Scale (CDRS) during the intravenous levodopa cycle from 0900 - 1500. The CDRS is a commonly utilized scale that is completed by an observer who judges the severity of LID (0-4) in 7 body parts (face, neck, trunk, both legs, and both arms) during as the subject performs the cognitive distraction task while standing on the force plate for 60 seconds. CDRS ratings are made every half hour during the LD dose cycle by the principal investigator (KC) or co-investigator.
Time Frame: Every half hour from 0900 to 1500
Measure: Count of Participants; unit: Participants
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
Number analyzed (Participants) | 28 | 16 | 35
Participants | 16 | 8 | 30
Statistical Analysis 1: Comparison: No Statin; Test type: Superiority; p = 0.011, Chi-squared; threshold for significance is 0.05, degrees of freedom = 2

4. Secondary Outcome: Clinical Dyskinesia Rating Scale (Peak)
Description: The Clinical Dyskinesia Rating Scale (CDRS) is a commonly utilized scale that is completed by an observer who judges the severity of Levodopa induced dyskinesia (LID) in 7 body parts (face, neck, trunk, both legs, and both arms) during the force plate stance with a cognitive distraction task for 60 seconds. All body parts are rated separately on this 0 (none) to 4 (severe - markedly impairs activities) scale. Thus, the total score can range from 0 - 28 with 28 indicating the most severe LID. Peak CDRS ratings are the 11:00 am ratings.
Time Frame: 11:00 am
Population: Historical use of a statin BEFORE beginning levodopa: excluded 2 participants that could not stand for 1 minute; No historical use of a statin: excluded 1 participant that had a pre-syncopal episode and was given time to recover before resuming ratings.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
Number analyzed (Participants) | 26 | 16 | 34
score on a scale | 1.9 (2.6) | 1.6 (2.8) | 3.6 (3.1)
Statistical Analysis 1: Comparison: No Statin; Test type: Superiority; p = 0.033, ANOVA; degrees of freedom = 75

ADVERSE EVENTS:
Time Frame: 3 months - time between the screening visit and completion of the day visit.
Description: Total # at risk for All Cause Mortality: 88 - Includes those withdrawn during the AE collection period.
  Total # at risk for SAE/AE: 80 - Excludes those withdrawn, did not complete day visit and therefore not at risk of AE during levodopa infusion/day visit.
Arm/Group | Statin Before Levodopa | Statin After Levodopa | No Statin
All-Cause Mortality (participants affected / at risk) | 1/32 | 1/17 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/16 | 3/35
Other Adverse Events (participants affected / at risk) | 0/29 | 1/16 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin Before Levodopa (N=29) | Statin After Levodopa (N=16) | No Statin (N=35)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin Before Levodopa (N=29) | Statin After Levodopa (N=16) | No Statin (N=35)
LightHeadedness (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Type II statins became more popular in use during the course of the study, which led to recruitment difficulties initially and a pivot to allowing most all statin drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04064294/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04064294/ICF_002.pdf